CLINICAL TRIAL: NCT06719310
Title: A Phase Ib/IIa, Randomized, Double Blinded, Perallel, Dosing Ranging, Placebo Controled and Proof of Concept Clinical Trial to Evaluate the Safety, Tolerability, PK and Antiviral Effect of ACC017 Tablet as Monotherapy/Combination With NRTI in Treatment naïve HIV-infected Adults
Brief Title: Phase Ib/IIa Clinical Study of ACC017 Tablets
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Aidea Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Chengdu Aidea Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADYY-ACC017-103&201
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded in the stage one, open in the stage two
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participant group 1 (Experimental): Stage one: ACC017 (Dose 1) Stage two: ACC017 (Dose 1)+FTC/TAF (200mg/25mg) QD
  Interventions: Drug: ACC017+FTC/TAF
- Participant group 2 (Experimental): Stage one: ACC017 (Dose 2) Stage two: ACC017 (Dose 2)+FTC/TAF (200mg/25mg) QD
  Interventions: Drug: ACC017+FTC/TAF
- Participant group 3 (Experimental): Stage one: ACC017 (Dose 3) Stage two: ACC017 (Dose 3)+FTC/TAF (200mg/25mg) QD
  Interventions: Drug: ACC017+FTC/TAF
- Participant group 4 (Placebo Comparator): Stage one: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACC017+FTC/TAF — ACC017+FTC/TAF
  Arms: Participant group 1; Participant group 2; Participant group 3
Drug: Placebo — Placebo
  Arms: Participant group 4

SUMMARY:
ACC017 is an integrase inhibitor that will be evaluated for the treatment of HIV infection. This phase Ib/IIa, randomized, double-blind, parallel, dose ranging, placebo-controlled 'proof of concept' study is designed to evaluate the safety, tolerability, pharmacokinetics and antiviral effect of ACC017 monotherapy and combined with FTC/TAF by sequency versus placebo in treatment-naïve HIV-1 infected adults. This study includes two stages, stage one is a single dose escalation, and all subjects will be co-administrated with FTC/TAF at 200 mg/25 mg on stage two. The study consists of a screening visit, baseline period, monotherapy period, and combination therapy period. Total 36 subjects will be randomized in a 5:1 ratio to receive one of three doses of ACC017 or placebo lasting for 10 days for monotherapy followed by 18 days for combination therapy.

DETAILED DESCRIPTION:
This phase Ib/IIa study in HIV-infected antiretroviral naive adult subjects is conducted to evaluate the safety, tolerability, pharmacokinetics and antiviral effect of ACC017 tablet as monotherapy/combination with NRTIs and to explore the recommended dose for the future pivotal clinical trial of ACC017. The study will be conducted as two stages. Stage one will includes a dose-ranging evaluation of ACC017 5mg, 40mg and 80mg once daily compared to placebo on the basis of safety, tolerability, pharmacokinetics and antiviral activity. Subjects will be randomized in a 5:1 ratio to receive one of three doses of ACC017 or placebo. Each subject will receive ACC017 tablet as monotherapy for 10 days and then followed by a combination with NRTIs for 18 days. In monotherapy, the enrolment into the next higher dose group will commence only when investigator and sponsor both agree that ACC017 is safe and well tolerated at a given dose. Stage two is open and subjects will continue to take ACC017 at the dose given on stage one in combination with FTC/TAF tablet at 200 mg/25 mg once daily for 18 days. Subjects randomized to receive placebo in stage one will receive the equivalent dose of ACC017 combined with FTC/TAF.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent and agree to comply to the study procedures and requests
2. Age range between 18 and 65 years old at the time of signing informed consent, regardless of gender
3. Body weight ≥40 kg, and BMI range between 18.5~29.9 kg/m2 (including the borderline) at screening
4. Documented HIIV-1 infection before screening, and never receive any antiHIV-1 drugs or vaccines after the diagnosis of HIV-1 infection
5. Agree not to use any antiviral drugs other than those allowed by protocol during study period.
6. Plasma HIV RNA≥5000 copies/mL at screening;
7. CD4+ T-lymphocyte count of >200 cells/μL

Exclusion Criteria:

1. Diagnosis of acute HIV infection at screening or unstable AIDS related disease within 4 weeks prior to screening.
2. Had PrEP and/or PEP treatment within 1 month prior to screening.
3. Had uncontrolled severe disease judged by investigator, such as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, NYHA class III or IV or fasting glucose ≥7.0 mmol/L.
4. History of serious allergy to drugs (such as aspirin or cephalosporin antibiotics) or their ingredients' or food (a fast, life-threatening systemic allergic reaction), or allergic disease requiring drug control (such as asthma, urticaria, atopic dermatitis [eczema].).
5. Any major gastrointestinal surgery (except uncomplicated appendectomy or cholecystectomy) or any surgery affecting drug absorption, distribution, metabolism and excretion within 6 months before screening; or possible elective surgery during the trial as judged by the investigator.
6. History of cancer(except cervical carcinoma in situ, or cutaneous basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ [Bowen's disease] that received radical surgery or treatment) within 5 years prior to screening.
7. Hb <90 g/L, or WBC count <1.5×109/L, or ANC count <0.6×109/L, or platelet count <50×109/L at screening.
8. ALT and/or AST > 2.5 times upper limit of normal (ULN), or TBIL > 1.5 × ULN, or DBIL > ULN, or ALB <30 g/L at screening.
9. SCr > 1.3 ×ULN, or Ccr <60 mL/min (Cockcroft-Gault formula) at screening,
10. Blood amylase or lipase >1.5 ×ULN
11. Subjects with a positive for HBsAg or anti-HCV, or those with anti-Tp positive who need to be treated required by investigator or their treatment period <7 days at screening.
12. Average smoked cigarettes more than 5 a day within 3 months prior to screening or unwilling to stop using any tobacco products during hospitalization.
13. Drinking more than 14 units per week within 3 months prior to screening ( 1 unit of alcohol is equivalent to 5% beer, 45 mL of 40% alcohol, 150mL of 12% alcohol), or a positive alcohol breath test at a screening or baseline visit, or unwilling to stop drink any alcohol-containing product during hospitalization.
14. Excessive consumption of tea, coffee or caffeine ( more than 8 cups per day on average, 1 cup of 250 mL) or unwilling to stop drinking tea, coffee, or caffeine during hospitalization.
15. Having taken pitaya, mango, grapefruit, star fruit or any preparations made from them, or food/drinking containing xanthine, caffeine or alcohol (e.g.chocolate, tea, coffee, cola and cocoa) or others that will affect the absorption, distribution, metabolism, excretion of drugs, within 48 hours prior to the first dose of experimental drugs, or unwilling to stop taking them during hospitalization.
16. Use of any potent or moderate CYP3A inhibitors (e.g. clarithromycin, thalimycin, ketocomazole, ketoconazole, itraconazole, and CYP3A4) or potent CYP3A4 inducers (e.g. rifampin, efavirenz,carbamazepine, phenobarbitone, phenytoin) within 14 days prior to the first dose of experimental drugs or within 5 half-lives(whichever is longer).
17. Use of any potent or moderate UGT1A inhibitors (e.g. silybin. Ritonavir) or potent UGT1A1 inducers (e.g. rifampin, carbamazepine) within 14 days prior to the first dose of experimental drugs or within 5 half-lives (whichever is longer).
18. Use of any prescription drug, nonprescription drug, Chinese traditional herbs within 14 days prior to the first dose of experimental drugs or within 5 half-lives (whichever is longer).
19. History of drug dependence (social, psychological and physical impairment due to excessive, impropriate or addictive use of substances for any non-medical reason) within 5 years prior to screening, or positive urine drug screen at screening or baseline.
20. Intolerance to venipuncture, or have a history of halo acupuncture or blood sickness, or have donated blood including component blood or have had substantial blood loss (more than 400 mL) or have received a blood transfusion within 3 months prior to screening, or plan to donate blood during study.
21. Have special dietary requirements at screening, or refuse to accept a standard diet.
22. Have participated in or are participating in another drug or medical device clinical study within 3 months prior to screening.
23. Women who are pregnant or breastfeeding or who have a positive blood pregnancy test at screening.
24. Have a birth plan (including conception, eggs or sperm donation) within 1 month before signing informed consent form until 3 months after last dose of experimental drugs or refuse to use effective any contraceptive methods.
25. Other conditions exist that, in the judgement of the investigator, make participation in this study unsuitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Report the incidence, severity and seriousness of adverse events, and the relationship between drug and AE | Day 1- Day 11
  Report the incidence, severity and seriousness of adverse events, and the relationship between drug and AE
HIV-1 RNA viral load change from baseline | Day 11
  HIV-1 RNA viral load change from baseline
Proportion of patients with HIV-1 RNA viral load <50 copies/mL | Day 29
  Proportion of patients with HIV-1 RNA viral load <50 copies/mL
Pharmacokinetics parameter: Cτ,ss | Day 10, Day 29
  Cτ,ss is defined as the steady-state plasma drug concentration at the end of the dosing interval after the last administration of a given dose on the monotherapy and combination therapy periods.
Pharmacokinetics parameter: Cmin,ss | Day 10
  Cmin,ss is defined as the minimum steady-state plasma drug concentration after the last dose of monotherapy.
Pharmacokinetics parameter: Cmax,ss | Day 10
  Cmax,ss is defined as the maximum steady-state plasma drug concentration after the last dose of monotherapy.
Pharmacokinetics parameter: AUC0-τ,ss | Day 1- Day 10
  AUC0-τ,ss is defined as the steady-state area under the plasma concentration-time curve from time zero to the any dosing interval of monotherapy.
Pharmacokinetics parameter: Tmax,ss | Day 1-Day 10
  Tmax,ss is defined as the time to reach steady-state maximum plasma concentration during monotherapy period.
Pharmacokinetics parameter: MRT0-τ,ss | Day 1-Day 10
  MRT0-τ,ss is defined as the steady-state mean residence time from time zero to any dosing interval of monotherapy.

SECONDARY OUTCOMES:
Changes over time in temperature of vital signs | Day 1-Day 29
  Temperature in degree Celsius.
Changes over time in pulse of vital signs | Day 1-Day 29
  Pulse in beat per minute.
Changes over time in systolic and diastolic blood pressure of vital signs | Day 1-Day 29
  Systolic and diastolic blood pressure in millimeters (mm) of mercury (Hg).
Changes over time in respiratory rate of vital signs | Day 1-Day 29
  Respiratory rate in breaths per minute.
Changes over time in heart rate as measured by electrocardiogram(ECG) | Day 1-Day 29
  Heart rate in beat per minute.
Changes over time in PR interval as measured by ECG | Day 1-Day 29
  PR interval is measured by ECG.
Changes over time in QRS duration | Day 1-Day 29
  QRS duration is measured by ECG.
Changes over time in QTc interval | Day 1-Day 29
  QTc interval is measured by ECG.
Changes over time in weight | Day 1-Day 29
  Weight is in kilograms.
Pharmacokinetics parameters: Cmax | Day 1-Day 2
  The maximum drug concentration following the first dose of monotherapy.
Pharmacokinetics parameters: Cτ | Day 2
  The drug concentration on the end of the first dosing interval of monotherapy.
Pharmacokinetics parameters: AUC0-τ | Day 2
  AUC0-τ is defined as the area under the plasma concentration-time curve from time zero to the first dosing interval of monotherapy.
Pharmacokinetics parameters: Tmax | Day 1- Day 2
  Time to reach the maximum drug concentration after the first dose of monotherapy.
Pharmacokinetics parameters: MRT0-τ | Day 1- Day 2
  MRT0-τ is defined as the steady-state mean residence time from time zero to the first dosing interval of monotherapy.
Report the incidence, severity and seriousness of adverse events, and the relationship between drug and AE | Day 11-Day 29
  Report the incidence, severity and seriousness of adverse events, and the relationship between drug and AE
HIV-1 RNA viral load changes from baseline over time | Day 2-Day 4, Day 8-Day 11, Day 21, Day 29
  HIV-1 RNA viral load changes from baseline over time
Proportion of patients with HIV-1 RNA viral load <50 copies/mL | Day 11
  Proportion of patients with HIV-1 RNA viral load <50 copies/mL
Proportion of patients with HIV-1 RNA viral load <200 copies/mL | Day 11, Day 29
  Proportion of patients with HIV-1 RNA viral load <200 copies/mL
The proportion of patients with HIV-1 RNA viral load <400 copies/mL | Day 11, Day 29
  The proportion of patients with HIV-1 RNA viral load <400 copies/mL
Changes in viral load from baseline to HIV-1 RNA viral load at nadir | Day 11
  Changes in viral load from baseline to HIV-1 RNA viral load at nadir
The proportion of nadir HIV-1 RNA <50 copies/mL | Day 11
  The proportion of nadir HIV-1 RNA <50 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Fujie, M.D., Ph.D., Principal Investigator — Beijing Ditan Hospital; Hu C Ying, Ph.D., Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, China